CLINICAL TRIAL: NCT05101707
Title: Combining taVNS With Early CIMT to Improve Health Outcomes of Infants With Unilateral Upper Extremity Weakness
Brief Title: CIMT and taVNS for Hemiplegia in Infants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Center of Neuromodulation for Rehabilitation (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 109558; P2CHD086844 (NIH)
Record Dates: First submitted 2021-10-01; First posted 2021-11-01 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Infant Development; Hemiplegia; Constraint Induced Movement Therapy
Keywords: transcutaneous auricular vagus nerve stimulation; constraint induced movement therapy; infant hemiplegia
MeSH Terms: conditions — Hemiplegia | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Intervention Model Description: CIMT plus taVNS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CIMT + taVNS (Experimental): The investigators will deliver taVNS paired with 40h of Constraint Induced Movement Therapy for unilateral weakness/hemiplegia
  Interventions: Device: transcutaneous auricular vagus nerve stimulation; Other: Constraint induced movement therapy

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — Applying a pulsed microcurrent to the auricular branch of the vagus nerve, timed with motor activity of the weaker arm/hand
  Other Names: taVNS
Other: Constraint induced movement therapy — Applying a custom-made splint constraint to the stronger hand/arm to encourage use of the weaker hand/arm in intensive therapy sessions
  Other Names: CIMT

SUMMARY:
Newborns who are born premature or suffer brain injury at birth are at risk for motor problems that may cause weakness in reaching and grasping on one side of the body. In older children, therapists may use a hand mitt and restraint for the stronger arm, to encourage use of the weaker side, called constraint-induced movement therapy (CIMT). Even with the high intensity therapy of CIMT, it typically takes between 40-120 hours total treatment time for most children to improve their motor skills. A non-invasive form of nerve stimulation, transcutaneous auricular vagus nerve stimulation (taVNS), stimulates a nerve by the ear that enhances learning motor skills. The purpose of this study is to evaluate the safety and effectiveness of taVNS to improve motor skills when paired with CIMT in infants with one-sided weakness at 6-18months of age.

DETAILED DESCRIPTION:
Recent pioneering studies have used neuromodulation combined with intensive motor therapies in adults after stroke. Few studies have investigated combining neuromodulation and evidence-based pediatric intensive therapies such as CIMT, and then only in older children with CP to enhance neuroplasticity and improve functional outcomes. The investigators are the first to use non-invasive transcutaneous auricular vagus nerve stimulation (taVNS) paired with a motor task of bottle-feeding in infants with feeding failure. taVNS paired with motor feeding activity was safe and over 50% infants attained full oral feeds who were slated to receive a gastrostomy tube (G-tube). With the unique collaboration of experts in brain stimulation, pediatric translational clinical science and pediatric occupational therapy in this pilot project, the investigators propose to expand the paradigm of pairing neuromodulation with motor training in at-risk infants by exploring the safety, feasibility, and effectiveness of delivering taVNS concurrently with CIMT. The hypothesis is that combining taVNS with intensive CIMT may boost neuroplasticity, allowing for delivery of infant therapy at a minimally effective dosage while improving infant outcomes.

The investigators aim to determine the feasibility and safety of taVNS in at-risk infants 6-18mo undergoing CIMT therapy in open label pilot trial and assess both infant tolerability and the therapist's ability to deliver high-quality CIMT along with taVNS.

ELIGIBILITY:
Inclusion Criteria:

Must have all of the following:

* 6-18 month-old infants with hemiplegia/motor asymmetry
* Must be able to participate in high intensity CIMT
* Gross Motor Function Classification System (GMFCS) level I-IV

Exclusion Criteria:

Must have none of the following:

* GMFCS level V
* severe motor impairment/quadriplegic involvement
* uncorrected blindness or deafness
* cardiomyopathy

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited participants from referrals from neonatal high risk development clinic, and referral from other rehab professionals seeing patients in their clinics from June 1, 2021 to July 30, 2024.
Pre-assignment Details: open label study without a washout period. all participants were receiving physical and occupational therapy for hemiplegia
Period: Overall Study
Arm/Group | CIMT + taVNS
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Open Label taVNS Paired With 40 Hours CIMT: infants with hemiplegia receive taVNs paired with constraint induced movement therapy for a total of 40h, 2h a day 5 days a week for 4 weeks
Arm/Group | Open Label taVNS Paired With 40 Hours CIMT
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: months of age] — months of age
  months of age | 16.7 [10 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: CIMT Fidelity
Description: Feasibility of delivering high fidelity CIMT therapy sessions while the therapist is also triggering taVNS using the Fidelity of Implementation Measure (FIRM) with scoring range (0-4), higher scores indicate greater consistency of therapy with established CIMT procedure
Time Frame: at 1 month
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Open Label taVNS Paired With 40 Hours CIMT
Number analyzed (Participants) | 3
score on a scale | 3.76 [3.58 to 3.76]

2. Primary Outcome: Quality of Upper Extremity Skills Test (QUEST), GRASP
Description: change in test of hand function and quality of movement between the right and left sides of the body, scoring range 0-100, higher scores indicate better hand function; from baseline to end of treatment
Time Frame: 1 month
Population: entire group (n=6) received 40h of CIMT with taVNS
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Open Label taVNS Paired With 40 Hours CIMT
Number analyzed (Participants) | 6
percentage of change from baseline | 209 (161)

3. Secondary Outcome: Gross Motor Function Measure-88 (GMFM-88)
Description: The Gross Motor Function Measure-88 (GMFM-88) assessment tool includes 88 items, each receiving a score from 0 to 3 (0 = does not initiate; 1 = initiates; 2 = partially completes; 3 = completes). Items span the spectrum of gross motor activities in five dimensions: A: Lying and Rolling (17 items), B: Sitting (20 items), C: Crawling and Kneeling (14 items), D: Standing (13 items), E: Walking, Running, Jumping (24 items). Every dimension score is expressed with a percentage. All dimension scores are then averaged to a total GMFM-88 percentage score, which is an estimate of the participant's gross motor function (0 = low motor function; 100 = high motor function).
Time Frame: 1 month
Population: entire group that received 40h of CIMT paired with taVNS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label taVNS Paired With 40 Hours CIMT
Number analyzed (Participants) | 6
units on a scale | 32 (28)

ADVERSE EVENTS:
Time Frame: 1 month
Description: recorded adverse events during sessions of taVNS-paired with CIMT
Arm/Group | CIMT + taVNS
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT05101707/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT05101707/ICF_000.pdf